CLINICAL TRIAL: NCT06256991
Title: Potassium Correction for Renin-angiotensin-aldosterone System Optimization in Chronic Kidney Disease
Brief Title: Potassium Correction for RAAS Optimization in Chronic Kidney Disease
Acronym: PROMISE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Amsterdam University Medical Center (Other); Frisius Medisch Centrum (Other); Isala (Other); Vifor Pharma, Inc. (Industry); Dutch Kidney Foundation (Other); Health Holland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 17237
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases; Hyperkalemia; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia; Hypertension | interventions — patiromer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, care providers and investigators will be blinded regarding the use of patiromer vs. placebo during the two study periods. Irbesartan will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patiromer (Experimental): All participants will receive patiromer 8.4g/d (powder for oral suspension) during one of the two 12-week study periods. Following a 6-week washout, participants will switch from the patiromer arm to the placebo arm or vice versa (cross-over design).
  Interventions: Drug: Patiromer 8400 MG [Veltassa]
- Placebo (Placebo Comparator): All participants will receive placebo 8.4g/d (powder for oral suspension) during one of the two 12-week study periods. Following a 6-week washout, participants will switch from the patiromer arm to the placebo arm or vice versa (cross-over design).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Patiromer 8400 MG [Veltassa] — Patiromer is a cation-exchanging polymer intended for oral intake that is not resorbed from the gastro-intestinal tract. Patiromer has been approved by the European Medicines Agency (EMA) and is available for clinical use in The Netherlands for the indication of hyperkalemia in adults. It contains calcium-sorbitol complex as a counter-ion. Patiromer increases the faecal excretion of potassium in the gastro-intestinal lumen by exchange with part of the calcium. This results in a lower concentration of free potassium in the gastro-intestinal lumen, reducing in turn plasma potassium concentration. After initiation of patiromer, a clinically significant reduction in plasma potassium can be observed at around 7 hours, the effect persists for approximately 24 hours. Patiromer is excreted by the fecal route, 24-48 hrs after ingestion. Since patiromer is not absorbed or metabolized by the body, other drugs are not expected to influence the efficacy of patiromer.
  Arms: Patiromer
Drug: Placebo — Placebo is a powder with a similar appearance, smell, and taste as patiromer, but without and clinically detectable effects. It is intended for oral intake.
  Arms: Placebo

SUMMARY:
The goal of this placebo-controlled, double-blinded cross-over trial is to test whether patiromer, compared with placebo, better enables up-titration of RAAS-blocker treatment in patients with chronic kidney disease stage 3b/4.

The main questions it aims to answer are:

* Does patiromer allow uptitration of irbesartan, resulting in a significant reduction in albuminuria and blood pressure?
* Does patiromer allow uptitration of irbesartan, resulting in a significant reduction in blood pressure?

The trial contains the following interventions:

* Participants will be switched from their ACEi/ARB to a standardised dose of irbesartan (150 mg/d).
* During two 12-week study periods, participants will receive either patiromer 8.4 g/d or placebo. The order of study periods is randomized.
* At the start of each study period irbesartan will be up-titrated to 300 mg/d.
* After 1 and 6 weeks, at both periods, plasma potassium will be measured and the irbesartan dose will be reduced to 150 mg/d in case plasma potassium exceeds 5.0 mmol/L.
* At 12 weeks from the start of the study period, the endpoints will be assessed.
* Between the two study periods, there is a 6-week washout. Irbesartan dose during the wash-out period will be 150mg/d. After washout, participants will switch from the patiromer arm to the placebo arm or vice versa.

DETAILED DESCRIPTION:
The PROMISE trial is a randomized, double-blind, placebo controlled cross-over trial where individuals are participating for 36 weeks. The trial consists of a 6-week run-in period, followed by two 12-week study periods, separated by a 6-week washout period.

First, during a run-in period, each participant will be converted from their ACEi/ARB dose to irbesartan 150 mg once daily. Individuals who already used irbesartan 150mg once daily before trial participation will remain on this dose during the run-in period. After six weeks, blood and 24-hour urine samples will be collected (baseline visit) and participants will be randomized to patiromer or placebo (start of study period A). The participant, research team, and treating physician will be blinded to treatment allocation (patiromer or placebo), while irbesartan will remain open-label.

At one week after start of study period A and B, participants will perform a home blood pressure measurement and visit a local lab to verify the plasma potassium level (safety visit), in combination with a scheduled phone consultation. The following actions may be taken: 1) If plasma potassium is >5.0 mmol/L or eGFR is >25% lower than baseline, the dose of irbesartan will be reduced to 150 mg/d and remain so during the remainder of the study period; 2) If systolic blood pressure is <110 mmHg, the participant has symptoms of hypotension, and plasma potassium is <5.0 mmol/L, antihypertensive co-medication may be adjusted, if applicable. If there is no antihypertensive co-medication that can be adjusted, the irbesartan dose will be reduced to 150 mg/d during the remainder of the study period.

At six weeks after start of the study period, there will be an in-hospital study visit. Blood samples will be collected, and office blood pressure will be measured. Any of the same two actions as described above may be taken in case of hyperkalaemia, severe acute kidney function decline or hypotension, respectively.

At the end of each 12-week study period, blood and 24-hour urine samples will be collected, and home (as well as office) blood pressure will be measured to establish the study endpoints. In addition, the study medication (patiromer/placebo) will be stopped and irbesartan dose will be reduced (or maintained) at 150 mg once daily. After a 6-week washout period, the second baseline will take place (measurements identical to the first baseline), which marks the start of study period B. During study period B, participants who had been randomized to patiromer in period A will now receive placebo and vice versa. The measurements during study period B will be identical to period A. At 12 weeks after the start of study period B, the protocol is completed and patients will return to their original medication.

The investigators chose a cross-over study design to be able to use participants as their own control; this will enhance statistical power and reduce the number of required participants. Based on previous studies, it is known that 6 weeks are sufficient to reach stable albuminuria and blood pressure after an ARB dose change. Therefore, even if halfway the 12-week study period a dose reduction is made, there is enough time for albuminuria and blood pressure to stabilize before the end of the study period (i.e., when the primary endpoint is established). A 6-week washout period is inserted to avoid carry-over effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* CKD stage 3b-4 (eGFR 15-44 mL/min/1.73 m2)
* Albumin-creatinine ratio >3 mg/mmol, or proteinuria >0.05g/24u, or protein-creatinine ratio > 5mg/mmol
* Systolic blood pressure >130 mmHg or use of one or more antihypertensive drugs;
* Serum K+ 4.0-5.0 mmol/L;
* On sub-maximal dose ACEi/ARB

Exclusion Criteria:

* prior ACEi/ARB dose reduction due to a drop in eGFR by >25% in the last year;
* history of severe hyperkalaemia (>6.0 mmol/L) in the last year;
* pregnancy or breastfeeding
* life expectancy <12 months
* the use of lithium, potassium-sparing diuretics, potassium supplements, trimethoprim or NSAIDS
* kidney transplant recipients, or diagnosis of autosomal dominant polycystic kidney disease or other non-glomerular kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Albumin-creatinine ratio (ACR) | At the end of both 12-week study periods (patiromer and placebo)
  The primary study endpoint is the difference in ACR in 24-hour urine at the end of each study visit, compared to the ACR at the start of the study period. This is a continuous variable that will be presented quantitatively. In case of non-normal distribution, this parameter will be log-transformed. The primary hypothesis test will be the difference between placebo and treatment groups after 2 periods.

SECONDARY OUTCOMES:
Blood pressure | At the end of both 12-week study periods (patiromer and placebo)
  Systolic and diastolic blood pressure, assessed by a 24-hour ambulatory blood pressure measurement at the end of each study period (continuous data)
Plasma potassium | At the end of both 12-week study periods (patiromer and placebo)
  Plasma potassium level at the end of each study period (continuous data)
Kidney function | At the end of both 12-week study periods (patiromer and placebo)
  Kidney function, as reflected by the estimated glomerular filtration rate (eGFR) using the combined cystatin C-creatinine-based CKD-EPI formula, at the end of each study period (continuous data)
Irbesartan dose | At the end of both 12-week study periods (patiromer and placebo)
  Irbesartan dose at the end of each study period (continuous data)
Adverse events | At the end of both 12-week study periods (patiromer and placebo)
  Numbers of AE/SAE during each study period (count data)

CONTACTS AND LOCATIONS:
Overall Officials: Liffert Vogt, prof. dr., Principal Investigator — Amsterdam University Medical Centre; Aaltje Adema, dr., Principal Investigator — Frisius Medisch Centrum; Femke Waanders, dr., Principal Investigator — Isala Zwolle; Martin de Borst, prof. dr., Study Chair — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Participants will be asked for permission to use collected personal information and biological samples for further research. Study data will be stored for 25 years in accordance with national guidelines.